CLINICAL TRIAL: NCT04043598
Title: Crystalloid Fluid Choice and Neurological Outcome in Patients After Subarachnoid Haemorrhage - a Multi-center Randomized Double-blind Clinical Trial
Brief Title: Crystalloid Fluid Choice and Neurological Outcome in Patients After Subarachnoid Haemorrhage
Acronym: CRYSTALLBrain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CRYSTALLBrain
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Subarachnoid Hemorrhage; Critical Illness; Infusion Fluid; Sodium Disorder
MeSH Terms: conditions — Subarachnoid Hemorrhage; Critical Illness | interventions — Sodium Chloride; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Multi-center investigator-initiated randomized-controlled double blind clinical trial comparing to already established treatment protocols.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high sodium infusion fluid (Active Comparator): Patients will exclusively receive 0.9% saline (sodium content 154mmol/l) for fluid maintenance and resuscitation from study inclusion until ICU/intermediate care (IMC) discharge.
  Interventions: Drug: 0.9% Sodium-chloride
- low sodium infusion fluid (Active Comparator): Patients will exclusively receive lactated Ringer's (sodium content 130mmol/l) for fluid maintenance and resuscitation from study inclusion until ICU/intermediate care (IMC) discharge.
  Interventions: Drug: Ringer's Lactate

INTERVENTIONS:
Drug: 0.9% Sodium-chloride — We will compare two already established treatment protocols: the use of normal saline versus lactated Ringer's for fluid therapy in patients with subarachnoid hemorrhage.
  Arms: high sodium infusion fluid
Drug: Ringer's Lactate — We will compare two already established treatment protocols: the use of normal saline versus lactated Ringer's for fluid therapy in patients with subarachnoid hemorrhage.
  Arms: low sodium infusion fluid

SUMMARY:
Patients with subarachnoid hemorrhage are prone to suffer from dysnatriemia. Evidence shows that hyponatriemia is associated with increased incidence of vasospasm, brain swelling and mortality in these patients. Patients with subarachnoid hemorrhage often require large amounts of iv fluids in order to maintain euvolemia and support cardiocirculatory function. Prior evidence shows that the type of infusion fluid significantly influences blood sodium content. Hence, this study evaluated whether the sodium content of the infusion solution impacts mortality and morbidity in patients with subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Background: Despite ongoing advances in critical care mortality and morbidity of patients with subarachnoid hemorrhage remains high. Secondary brain injuries related to cerebral vasospasm and consecutive ischemic brain injury and intracerebral edema are the main contributors to mortality and morbidity in these patients. Evidence points towards low serum sodium levels being one of the significant risk factors for of secondary brain injury in this population. Previous studies show that fluid resuscitation with normal saline results in higher serum sodium levels and higher serum osmolality when compared to balanced infusates in patients with subarachnoid hemorrhage.

Aim: The primary objective of this study is to evaluate whether the use of a sodium-rich infusion (normal saline) results in better clinical outcome when compared to a sodium-depleted infusion (lactated Ringer's) in patients with subarachnoid hemorrhage. The primary endpoint will be the occurrence of clinically relevant vasospasm requiring immediate treatment. In addition, the investigators will assess other relevant complications such as long and short-term mortality, significant brain edema requiring conservative therapy or/and operative hemicraniectomy, as well as further patient-relevant outcomes such as days on organ support, postoperative infections, length of stay and long-term disability/mortality.

Study intervention: All patients admitted to a participating hospital with the diagnosis of intracerebral bleeding will be screened and if eligible, randomized to one of the study arms. Individual patient's consent will be sought. Thereafter, patients will receive only the allocated study fluid for fluid maintenance and resuscitation from study inclusion until ICU/intermediate care (IMC) discharge. Neurological evaluation will be performed hourly for the initial phase and thereafter two hourly. Serum sodium, osmolality, fluid, water and electrolyte balance as well as acid-base homeostasis will be evaluated daily. Further, specific assessment of renal, cardiac and immune function takes place at 5 pre-specified time-points (day 1,3,7,10 and at ICU/IMC discharge).

After ICU/IMC discharge patients will be followed for evaluation of secondary endpoints. Long-term disability will be assessed by telephone interview based on the modified the Rankin-Scale and the Glasgow Outcome Scale Extended.

Sample Size: Sample size calculation was based upon the investigators' ICU's registry data. In 2017, 44.38% patients with subarachnoid hemorrhage reached the predefined endpoint of clinically relevant vasospasm requiring immediate intervention. A clinically relevant effect size was determined to be an improvement in outcome of 15%. Based on these results a patient number of n = 160 for each group was determined under estimation of a 15% drop out rate.

ELIGIBILITY:
Inclusion Criteria:

All adult patients suffering from non-traumatic subarachnoid haemorrhage.

Exclusion Criteria:

* Patients with major intra-cranial trauma
* Diagnosis of an AV-malformation as the source of subarachnoid hemorrhage on the primary CT/MRI or angiography
* More than 24 hours after diagnosis of subarachnoid haemorrhage as diagnosed by cerebral imaging (CT scan or MRI)
* Patients with clear limitation to therapy at hospital admission (eg ICU admission for evaluation of organ donation)
* Declining of informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with clinically relevant vasospasms | From ICU admission until discharge (usually within the first 21 days)
  Defined as new neurologic deficit requiring immediate intervention

SECONDARY OUTCOMES:
Number of ICU deaths | From ICU admission until discharge (usually within the first 21 days)
  Death on the ICU
Number of In-hospital deaths | From hospital admission to hospital discharge (usually within the first 21 days)
  Death during hospital stay
Number of severe vasospasms requiring endovascular treatment | From hospital admission to hospital discharge (usually within the first 21 days)
  Number of severe vasospasms requiring endovascular treatment
Number of patients needing decompressive hemicraniectomy | From hospital admission to hospital discharge (usually within the first 21 days)
  Operative intervention needed for high intracranial pressure
Difference in modified RankingScale | At day 90 and 180
  Scale ranges from 0-5 (0 = no symptoms; 5= severe disability)
Difference in Glasgow Outcome Scale | At day 90 and 180
  Scale ranges from 1-8 (1 is dead 7 good recovery)
Difference in mini Montreal Cognitive Assessment | At day 90 and 180
  Max score depends on age and education (the higher the score the better the cognition)
Difference in Long-term mortality | At day 90 and 180
  Death at 90 and 180 day
Length of stay | ICU stay and hospital stay (usually between 1-30days)
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Messmer, MD, Principal Investigator — Department of Intensive Care, Inselspital, Bern University Hospital and University of Bern, Bern, Switzerland
Locations (3):
- Switzerland (3):
  - Department of perioperative Intensive Care Medicine, Sankt Gallen, Canton of St. Gallen
  - Department of Intensive Care, Bern University Hospital and University of Bern, Bern, Switzerland, Bern
  - Department of Intensive Care Medicine, Geneva

IPD SHARING:
Plan to Share IPD: No
Information will be available upon request.

REFERENCES:
- [Background] Messmer AS, Pitteloud M, Quintard H, Pietsch U, Muller M, Filipovic M, Jakob SM, Z'Graggen WJ, Schefold JC, Pfortmueller CA. CRYSTALLBrain: crystalloid fluid choice and neurological outcome in patients with non-traumatic subarachnoid haemorrhage-a study protocol for a multi-centre randomised double-blind clinical trial. Trials. 2025 Oct 17;26(1):422. doi: 10.1186/s13063-025-09099-9. PMID 41107997